CLINICAL TRIAL: NCT06752018
Title: Inflammation: a Key Contributor to Heart Disease and Diabetes?
Brief Title: Inflammation's Impact on Heart Disease and Diabetes
Acronym: INFO
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-91-24
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-12

CONDITIONS: Inflammation; Obesity and Type 2 Diabetes; Obesity; Metabolic Syndrome; Anti-Inflammatory Agents
Keywords: Disease; Overweight; overnutrition; body weight; Insulin resistance; Inflammation; Anti-Inflammatory Agents
MeSH Terms: conditions — Inflammation; Obesity; Diabetes Mellitus, Type 2; Metabolic Syndrome; Disease; Overweight; Overnutrition; Body Weight; Insulin Resistance | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Omental adipose tissue
  * Subcutaneous adipose tissue
  * Whole blood
  * Plasma
  * Serum
  * Feces
  * Saliva
  * Liver
  * Intestine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Obese gastric bypass patients
  Interventions: Procedure: Gastric bypass
- Lean healthy controls

INTERVENTIONS:
Procedure: Gastric bypass — Roux-en-Y gastric bypass or sleeve gastrectomy
  Groups: Obese gastric bypass patients

SUMMARY:
The goal of this observational study is to evaluate the inflammatory response associated with cardiometabolic diseases, and whether these can be reduced by ex vivo treatment with therapeutic agents. Briefly, the study involves two populations: healthy volunteers and severely obese patients undergoing weight-loss surgery. The main questions the study seeks to address are:

1. To investigate if the therapeutic agents modulate the inflammatory response linked to obesity and cardiometabolic disease?
2. What underlying factors contribute to variations in individual responses?

Researchers will examine differences between healthy participants and those undergoing weight-loss surgery to assess the potential impact of weight loss on responsiveness and overall outcomes.

Participants will:

* Undergo initial testing to evaluate their baseline response.
* Provide samples during surgery for further analysis.
* Participate in follow-up assessments to track changes over time.

DETAILED DESCRIPTION:
The goal of this observational study is to investigate the relationship between treatment responsiveness and inflammation both systemically in blood, and peripherally in tissue biopsies, focusing on its relevance to cardiometabolic disease and associated conditions. The study aims to develop a predictive model to identify individuals most likely to benefit from anti-inflammatory treatments, thus supporting personalized therapeutic strategies.

Main research questions:

1. To investigate if the therapeutic agents modulate the inflammatory response linked to obesity and cardiometabolic disease
2. To determine the underlying factors that contribute to variations in individual responses to anti-inflammatory drugs

Study design:

The study will involve two participant groups:

* Healthy control group, composedrised of normal weight individuals
* Obese adult patients, scheduled to undergo bariatric surgery.

Participant procedures:

* Baseline testing: An initial test will evaluate treatment responsiveness.
* Tissue sampling: Tissue biopsies are obtained during surgery and undergo detailed analyses, including ex vivo treatments
* Follow-up assessments: Participants will be reassessed a year after surgery to evaluate long-term outcomes.

Methods:

* Molecular studies: Whole blood and peripheral tissue biopsies (adipose tissue, liver, muscle and intestinal biopsies) will be analyzed to identify cellular and molecular pathways associated with treatment responsiveness.
* Predictive modeling: Clinical, molecular, and biochemical data will be integrated to create a model predicting individual responsiveness.
* Insulin sensitivity analysis: Advanced imaging techniques will measure tissue-specific glucose uptake.

Hypotheses: Impaired ability to regulate the inflammatory response correlates with cardiometabolic disease.

Anticipated Outcomes:

The study seeks to support precision medicine approaches for addressing cardiometabolic disease.

This research builds on previous findings about the role of inflammation in cardiometabolic dysfunction. By differentiating responders from non-responders, the study aims to support targeted therapeutic strategies for inflammation and cardiometabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Individuals willing and able to give appropriate oral and written informed consent
* Men and women over 18 years of age.
* Correct body mass index (BMI) (Lean controls: 18.5-24.9 kg/m2. Obese gastric bypass patients: 35-50 kg/m2)

Exclusion Criteria:

* The individual does not follow instructions given in the research study.
* Pregnancy.
* Significant gastrointestinal problems.
* Use of tobacco.
* The individual consumed alcohol within two days prior to the study visit
* Active cancer within 5 years.
* Use of dietary supplements that impact the inflammatory resolution process (e.g., fish oils), and the person is not willing to discontinue the use of the supplements 1 week prior to the visits.
* Underlying cardiometabolic disease, or medication related to such disease (e.g., blood pressure medication, insulin to treat diabetes, etc.).
* Underlying inflammatory disease, or medication related to such disease.
* The individual states that they have increased bleeding tendency or are using anti-coagulant (blood-thinning) medication.
* For obese patients only: The individual has lost more than 8% of his/her body weight since their clinical referral for surgery or has lost more than 3% of his/her body weight in the 4 months leading up to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy controls and obese patients, scheduled to undergo bariatric surgery without a pre-surgical diet
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Whole blood ROS prooduction | At baseline and 1 year post surgery
  The primary endpoint of the study is the therapeutic agent-induced reduction in reactive oxygen species (ROS) production in whole blood, following stimulation with N-Formylmethionyl-leucyl-phenylalanine (fMLP), escherichia coli (E. coli), and phorbol myristate acetate (PMA).
Whole blood ROS production | At the time of enrollment
  The primary endpoint of the study is the therapeutic agent-induced reduction in ROS production in whole blood, following stimulation with fMPL, E. coli, or PMA

CONTACTS AND LOCATIONS:
Overall Officials: Emma Börgeson, Dr., PhD, MSc, Principal Investigator — University of Aarhus
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided